CLINICAL TRIAL: NCT01948596
Title: The Synchronized Trial on Expectant Mothers With Depressive Symptoms by Omega-3 PUFAs (SYNCHRO) : Open Trial
Brief Title: The Synchronized Trial on Expectant Mothers With Depressive Symptoms by Omega-3 PUFAs (SYNCHRO): Open Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tokyo Medical University (Other)
Collaborators: China Medical University, Taiwan (Other); Japan Society for the Promotion of Science (JSPS) (Unknown); University of Toyama (Other); Chiba University (Other)
Responsible Party: Principal Investigator, Daisuke Nishi, Assistant Professor, Tokyo Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYNCHRO-Open
Record Dates: First submitted 2013-09-12; First posted 2013-09-23 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Pregnancy; Depression
Keywords: pregnant women; depression; depressive symptoms; omega-3 fatty acids
MeSH Terms: conditions — Depression | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omega-3 polyunsaturated fatty acids (Experimental): 1200mg eicosapentaenoic acid (EPA) and 600mg docosahexaenoic acid (DHA) daily
  Interventions: Dietary Supplement: Omega-3 polyunsaturated fatty acids

INTERVENTIONS:
Dietary Supplement: Omega-3 polyunsaturated fatty acids
  Other Names: 1200mg EPA and 600mg DHA daily

SUMMARY:
The present study aims to examine the efficacy and safety of omega-3 polyunsaturated fatty acids for pregnant women with depressive symptoms.

DETAILED DESCRIPTION:
Maternal depression can have a significant harmful influence on both mothers and children. Considering the possibility of adverse effects of antidepressants and previous meta-analyses showing the positive effects of omega-3 polyunsaturated fatty acids (PUFAs) supplementation in reducing depressive symptoms, omega-3 PUFAs may provide a safe strategy. The investigators evaluate efficacy and safety of omega-3 PUFAs for pregnant women with depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant women aged 20 years or older
2. between 12-24 weeks gestation
3. a Japanese conversational ability in Japan site or a Mandarin conversational ability in Taiwan site to understand the scope of the present trial and to provide written consent for study participation
4. planned to return to the hospital for checkup at 4-6 weeks after childbirth
5. an Edinburgh Postnatal Depression Scale (EPDS) score is 9 or more
6. to have good physical health judged by obstetricians.

Exclusion Criteria:

1. history and current suspicion of psychosis or bipolar I disorder or substance-related disorder or eating disorder or personality disorder
2. the item of EPDS concerning suicide ideation is 2 or more
3. other serious psychiatric symptoms such as self-harm behavior or in need of rapid psychiatric treatment
4. difficult to expect a normal birth (ex: fetal malformation etc.)
5. having a history of bleeding disorder such as von Willebrand's Disease
6. regular treatment with aspirin or warfarin within the last 3 months
7. a smoking habit of ≥40 cigarettes per day
8. regular treatment with ethyl icosapentate or regular consumption of omega-3 PUFA supplements within the last 3 months
9. a habit of eating fish ≥4 times per week.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
total score of the Hamilton Rating Scale for Depression (HAMD) | Twelve weeks

SECONDARY OUTCOMES:
total score of HAMD | 4-6 weeks after childbirth
total scores on the Edinburgh Postnatal Depression Scale (EPDS) | Twelve weeks, 4-6 weeks after childbirth
total score of the Beck Depression Inventory Ⅱ(BDI-Ⅱ) | Twelve weeks, 4-6 weeks after childbirth
major depressive disorder (MDD) as determined by the depression module of the Mini International Neuropsychiatric Interview (MINI) | Twelve weeks, 4-6 weeks after childbirth
omega-3 fatty acids concentrations in erythrocytes | Tweve weeks, 4-6 weeks after childbirth
brain-derived neurotrophic factor (BDNF) in serum | Twelve weeks, 4-6 weeks after childbirth
IF-6 in plasma | twelve weeks, 4-6 weeks after childbirth
oxytocin in plasma | twelve weeks, 4-6 weeks after childbirth
TNF-alpha in plasma | twelve weeks, 4-6 weeks after childbirth
IL-1 beta in plasma | twelve weeks, 4-6 weeks after childbirth
phospholipase A2 in plasma | twelve weeks, 4-6 weeks after childbirth

OTHER OUTCOMES:
gestational age | at childbirth
gestational diabetes mellitus | 4-6 weeks after childbirth
gestational hypertension or preeclampsia | 4-6 weeks after childbirth
induced labour | at childbirth
estimated blood loss | at childbirth
cesarean section | at childbirth
operative vaginal delivery | at childbirth
birthweight | at childbirth
one minute apgar | 4-6 weeks after childbirth
5-minute apgar | 4-6 weeks after childbirth
neonatal intensive care unit admission | 4-6 weeks after childbirth
cholesterol | twelve weeks and 4-6 weeks after childbirth

CONTACTS AND LOCATIONS:
Overall Officials: Daisuke Nishi, M.D., Ph.D., Principal Investigator — Tokyo Medical University; Kuan-Pin Su, M.D., Ph.D., Principal Investigator — China Medical Univeristy
Locations (3):
- Japan (2):
  - Toda Maternity Hospital, Toda, Saitama
  - Tokyo Medical University, Shinjuku-ku, Tokyo
- China Medical University, Taichung, Taiwan

REFERENCES:
- [Result] Nishi D, Su KP, Usuda K, Chiang YJ, Guu TW, Hamazaki K, Nakaya N, Sone T, Sano Y, Ito H, Isaka K, Hashimoto K, Hamazaki T, Matsuoka YJ. Omega-3 fatty acid supplementation for expectant mothers with depressive symptoms in Japan and Taiwan: An open-label trial. Psychiatry Clin Neurosci. 2016 Jun;70(6):253-4. doi: 10.1111/pcn.12388. Epub 2016 May 6. No abstract available. PMID 27004997
- [Derived] Nishi D, Su KP, Usuda K, Chang JP, Chiang YJ, Guu TW, Hamazaki K, Nakaya N, Sone T, Hashimoto K, Hamazaki T, Matsuoka YJ. Differences between Japan and Taiwan in the treatment of pregnant women with depressive symptoms by omega-3 fatty acids: An open-label pilot study. Nutr Neurosci. 2019 Jan;22(1):63-71. doi: 10.1080/1028415X.2017.1354540. Epub 2017 Jul 28. PMID 28752805